CLINICAL TRIAL: NCT03940443
Title: Differences in Mortality and Morbidity in Patients Suffering a Time-critical Condition Between Ground Emergency Medical Services and Helicopter Emergency Medical Services - a Descriptive and Comparative Study
Brief Title: Differences in Mortality and Morbidity in Patients Suffering a Time-critical Condition Between GEMS and HEMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, David Summermatter, Principal Investigator, Dalarna County Council, Sweden
Other Study IDs: HDa 5.2.2-2017/745
Record Dates: First submitted 2019-03-13; First posted 2019-05-07 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Ambulances; Traumatic Brain Injury; Acute Myocardial Infarction
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ground Emergency Medical Services: Patients suffering TBI or acute MI and has been treated by GEMS dispatched by an emergency dispatch centre.

SUMMARY:
Introduction: Patients suffering a time-critical medical condition require rapid prehospital assessment and treatment and most often quick transportation to definitive care. This can be decisive for patient outcome. In order to minimize time from assessment to treatment, thus lowering mortality and morbidity, it is important to have a well-coordinated chain of care. The efficient use of Ground Emergency Medical Services (GEMS) and Helicopter Emergency Medical Services (HEMS) is essential in such a chain of care.

Objectives: The aim is to describe differences in mortality, morbidity, assessment and treatment of two time-critical conditions, traumatic brain injury (TBI) and acute myocardial infarction (MI), in patients assessed by GEMS and HEMS respectively.

Method: The project consists of a descriptive observational study and comparative cohort study. Inclusion criteria are patients considered to be suffering from TBI and acute MI, which are treated by GEMS or HEMS in the regions of Uppsala, Jämtland/Härjedalen, Dalarna and Värmland.

Clinical significance: The results expect to be the basis for further studies aiming to optimize the utilization of GEMS and HEMS.

DETAILED DESCRIPTION:
Background Efficient healthcare can be decisive for patients who suffer an out-of-hospital time-critical medical condition. If untreated these conditions can compromise health and even become life-threatening. The most common time-critical conditions assessed and treated in the prehospital environment are cardiac arrest, chest pain, stroke, severe respiratory difficulties and severe trauma. In addition to receiving rapid assessment and immediate treatment, it is also important that these patients are quickly transported to a location where they can receive the appropriate level of care.

If a person is suffering from an out-of-hospital time-critical medical condition, the emergency medical dispatch center is alerted when contacted by the use of '112' the emergency phone number common to European countries. An operator will answer the call and assess the situation using a medical criteria-based index . The operator will than dispatch the right resource, either Ground Emergency Medical Services (GEMS) or Helicopter Emergency Medical Services (HEMS).

The dispatching of HEMS has long been considered as a weak link in the chain of response. The use of HEMS is region specific and that the mechanism of injury is a poor predictor for HEMS dispatch. Dispatch criteria should be designed to match specific systems.

The prehospital care in Sweden has developed rapidly over recent decades. Prehospital care today is a system in which qualified prehospital care providers deliver advanced emergency healthcare. GEMS vehicles are staffed with at least one registered nurse (RN) and over the years programs has been developed, which leads to at postgraduate diploma in prehospital care nursing. GEMS has less access to medical-technical equipment for advanced medical life support and critical care. The HEMS medical staff consists of a RN with a postgraduate diploma in prehospital care nursing and a physician, specialized in anaesthesia and intensive care and HEMS is equipped for advanced life support and critical care interventions. All of Sweden´s Emergency Medical Services (EMS) organisations require educational programs and certification for prehospital trauma and emergency medical care on a yearly basis. These educational programs aim to improve emergency care based on evidence based medicine. Previous studies have demonstrated that EMS provides rapid access to the healthcare system, quality care on scene, and transport with support en-route to appropriate care if not provided on scene. An increased survival rate could be identified in trauma patients if transported by HEMS, compared to GEMS. Another study reported increased survival rate of patients over 55 years of age who suffered minor trauma and where transported by HEMS compared to GEMS. Previous studies has also shown an advantage in using HEMS in treating patients with acute MI, initiating treatment as early as possible. The time gained, using HEMS, in treating acute MI was reported to reduced mortality compared to patients treated by GEMS.

There is a steadily growing body of literature that describes the activities in both GEMS and HEMS and the assessment and treatment of Traumatic Brain Injury (TBI) and acute Myocardial Infarction (MI). But these studies are not generalisable to the Swedish prehospital environment, due to the importance of evaluating triage criteria for HEMS activation by local and regional authorities and the variation of health care system in which GEMS and HEMS operate. A systematic collection and analysis of incidence and outcomes in prehospital care of time-critical conditions can therefore increase dispatch accuracy and contribute to knowledge about which patients should be assessed and treated by GEMS and HEMS, respectively. This, in turn can lead to cost-effectiveness and better outcomes. Previous studies have been criticized for the low quality of evidence and variation in study methods, which overall has resulted in a lack of credibility in the conclusions of the studies.

TBI is a major cause of death, disability and cost to society. The perceived benefit of HEMS transport of trauma patients, including TBI is driven by the principle that time is a critical factor in the survival of severely injured patients. For patients with acute MI, time to treatment should be short as possible because every delay increases mortality. Since today, from a national perspective, both descriptive data and evidence in the form of studies comparing GEMS and HEMS are modest, it is very important to describe GEMS and HEMS for assessment, treatment and outcome of patients suffering from TBI and acute MI. Once a thorough description of GEMS and HEMS has been completed, hypothesis-generating controlled studies can be initiated. The project is expected to contribute to optimisation of the prehospital assessment and treatment of TBI and acute MI and the role of GEMS and HEMS in Sweden.

Overall aim To describe and to compare morbidity and mortality, assessment and treatment of TBI and acute MI in patients treated by GEMS and HEMS.

Specific aim Study I To describe the scope and characteristics of GEMS and HEMS assessing and treating patients with TBI and acute MI in the field of prehospital care and to illustrate the complexity of the topic. The collected data will be the starting point for study II.

Study II To understand the effects of GEMS compared to HEMS in patients suffering from TBI and acute MI and what care logistics should we use. Previous collected data from study I will be used for this purpose.

Research questions

Study I

1. What is the incidence of mortality and morbidity in the assessment and treatment of TBI and acute MI of GEMS and HEMS?
2. What types of assessment and treatment are performed in patients with TBI and acute MI?

Study II

1. What are the field diagnosis accuracy related to final diagnosis? Are there differences in diagnose accuracy in patients treated and transported with GEMS vs. HEMS?
2. What are the differences between GEMS vs. HEMS on mortality and morbidity in patients suffering from TBI and acute MI?

Hypothesis (study II): HEMS compared to GEMS provides significant time gains resulting in fewer morbidity and reduced mortality when assessing and treating patients with TBI and acute MI.

Design: Study I is a descriptive observation study with quantitative approach. Study II consists of a comparative cohort study with 30-day follow up. These studies will be reported according to STROBE´s recommendations for observational studies and cohort studies. The project will be registered in ClinicalTrials.gov before the start of the study.

Setting

Population:

Study I consists of patients considered to be suffering a TBI or acute MI and been treated by either GEMS or HEMS during the period of January 1st, 2018 to December 31st, 2018. Inclusion criteria are GEMS and HEMS prehospital care providers, men and women ≥18 years of age in a time-critical condition. Exclusion criteria are men and women < 18 years of age in a non-time-critical condition. Participating counties are located in the middle of Sweden.

Study II consists of patients considered to be suffering from a TBI or acute MI treated by GEMS prehospital care providers (Reference) (n=2000) and HEMS (Exposed) (n=2000) during the period of January 1st, 2017 to December 31st, 2018. Inclusion criteria are GEMS and HEMS prehospital care providers, men and women ≥18 years of age in a time-critical condition. Exclusion criteria are men and women < 18 years of age. Participating counties are located in the middle of Sweden.

Data collection Data for both studies is collected from existing digital and manual prehospital care reports (digital models: Cosmic, Ortivus, Paratus, TakeCare and manually written prehospital care reports (PCR)). The participating prehospital care providers will be the regional council of Uppsala, Jämtland/Härjedalen and Dalarna and the county council of Värmland. Data retrieved is scene location, time from dispatch to arrival to the patient on scene, time from dispatch to prehospital assessment/treatment, time from dispatch to patient arrival at the receiving health care facility, location of the receiving facility, type of condition, vital signs in the prehospital setting, treatment and survey of the patient. Searching and extracting data will be done using protocols where the study outcomes are documented as intended to answer the purpose of the study. Exported data from all patient record systems are reviewed for quality.

The IBM SPSS Version 25 Statistics Program will be used. The collected data will be processed with descriptive and comparative analyses as with regression models to evaluate the significance of variables for medical complications and mortality.

Exposed group: Patients suffering TBI or acute MI and has been treated by HEMS crews dispatched by an emergency dispatch centre re in all the counties.

Reference group: Patients suffering TBI or acute MI and has been treated by GEMS dispatched by an emergency dispatch centre.

Possible confounders Several confounders are yet unknown but this will be probably clarified by study I.

Outcome The primary outcome is mortality, and will be controlled with measure of time from dispatch to assessment and treatment to patient arrival at the receiving medical facility The secondary outcomes are comorbidity (diabetes), medical complications (Infection, haemorrhage) and 30-day mortality. Independent variables: HEMS vs GEMS and these groups will be controlled for age, sex and possible other variables that will be examined for their impact on regression models

Description of the groups (Study II) Exposed group: Patients suffering TBI or acute MI and has been treated by helicopter emergency medical service crews dispatched by an emergency dispatch center.

Reference group: Patients suffering TBI or acute MI and has been treated by ground emergency medical service care providers dispatched by an emergency dispatch center.

Power calculation: A power calculation is made in study II where comparative analysis are to be used.

Description of project logistics Information on the aim of study I and its implementation will be provided to the staff at all HEMS bases and to all ambulance stations in the regions participating in the study. The information will be given primarily to the medical director and the director of operations responsible for HEMS operations and GEMS. Data extract from digital PCR systems will be carried out by the operation managers. Manual data collection from HEMS is carried out by the collaborator of the study on the basis of approval from the director of operations. Data extracts of patients considered to suffer an TBI or acute MI are performed based on the outcomes of the study. Data extracts are handed over unidentified to researcher and is provided in a pre-defined folder on the computer of the responsible researcher through the server of the region where the computer is encrypted.

ELIGIBILITY:
Inclusion Criteria:

Patients suffering from a time-critical condition:

* Cardiac arrest
* Acute myocardial infarction
* Severe chest pain
* Stroke
* Severe respiratory difficulties
* Severe trauma

Exclusion Criteria:

Patient in a non time-critical condition:

* Minor trauma
* Minor respiratory difficulties
* Minor chest pain
* Minor neurologic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients considered to be suffering a TBI or acute MI and been treated by either GEMS or HEMS.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Mortality | January 1st, 2017 to December 31st, 2018
  The primary outcome is mortality, and will be controlled with measure of time from dispatch to assessment and treatment to patient arrival at the receiving medical facility. Timeframe from inclusion until death, up to 30 days. The outcome will be reported in numbers by proportion of participants and with tables in percentage.

OTHER OUTCOMES:
Comorbidity | January 1st, 2017 to December 31st, 2018
  The secondary outcomes are comorbidity (diabetes), medical complications (Infection, haemorrhage). Timeframe from inclusion until death, up to 30 days. The outcome will be reported in numbers by proportion of participants and with tables in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: David Summermatter, RN, Principal Investigator — Dalarna County Coucil
Locations (1):
- Region Dalarna, Falun, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krafft T, Garcia Castrillo-Riesgo L, Edwards S, Fischer M, Overton J, Robertson-Steel I, Konig A. European Emergency Data Project (EED Project): EMS data-based health surveillance system. Eur J Public Health. 2003 Sep;13(3 Suppl):85-90. doi: 10.1093/eurpub/13.suppl_1.85. PMID 14533755
- [Background] Georgette E, Simon B, James R. HEMS dispatch: A systematic review. Trauma. 2018;20(1):8.
- [Background] Suserud B-O, Lundberg L. Prehospital akutsjukvård. 2 ed. Stockholm: Liber; 2016. 560 p.
- [Background] Delgado MK, Staudenmayer KL, Wang NE, Spain DA, Weir S, Owens DK, Goldhaber-Fiebert JD. Cost-effectiveness of helicopter versus ground emergency medical services for trauma scene transport in the United States. Ann Emerg Med. 2013 Oct;62(4):351-364.e19. doi: 10.1016/j.annemergmed.2013.02.025. Epub 2013 Apr 9. PMID 23582619
- [Background] Andruszkow H, Hildebrand F, Lefering R, Pape HC, Hoffmann R, Schweigkofler U. Ten years of helicopter emergency medical services in Germany: do we still need the helicopter rescue in multiple traumatised patients? Injury. 2014 Oct;45 Suppl 3:S53-8. doi: 10.1016/j.injury.2014.08.018. PMID 25284235
- [Background] Andruszkow H, Schweigkofler U, Lefering R, Frey M, Horst K, Pfeifer R, Beckers SK, Pape HC, Hildebrand F. Impact of Helicopter Emergency Medical Service in Traumatized Patients: Which Patient Benefits Most? PLoS One. 2016 Jan 15;11(1):e0146897. doi: 10.1371/journal.pone.0146897. eCollection 2016. PMID 26771462
- [Background] Blankenship JC, Haldis TA, Wood GC, Skelding KA, Scott T, Menapace FJ. Rapid triage and transport of patients with ST-elevation myocardial infarction for percutaneous coronary intervention in a rural health system. Am J Cardiol. 2007 Sep 15;100(6):944-8. doi: 10.1016/j.amjcard.2007.04.031. Epub 2007 Jul 2. PMID 17826374
- [Background] Hesselfeldt R, Pedersen F, Steinmetz J, Vestergaard L, Simonsen L, Jorgensen E, Clemmensen P, Rasmussen LS. Implementation of a physician-staffed helicopter: impact on time to primary PCI. EuroIntervention. 2013 Aug 22;9(4):477-83. doi: 10.4244/EIJV9I4A77. PMID 23965353
- [Background] Pathan SA, Soulek J, Qureshi I, Werman H, Reimer A, Brunko MW, et al. Helicopter EMS and rapid transport for ST-elevation myocardial infarction: The HEARTS study. Journal of Emergency Medicine, Trauma and Acute Care. 2017;2017(1):8.
- [Background] Thomas SH, Blumen I. Helicopter Emergency Medical Services Literature 2014 to 2016: Lessons and Perspectives, Part 1-Helicopter Transport for Trauma. Air Med J. 2018 Jan-Feb;37(1):54-63. doi: 10.1016/j.amj.2017.10.006. Epub 2017 Dec 6. No abstract available. PMID 29332779
- [Background] Thomas SH, Blumen I. Helicopter Emergency Medical Services Literature 2014 to 2016: Lessons and Perspectives, Part 2-Nontrauma Transports and General Issues. Air Med J. 2018 Mar-Apr;37(2):126-130. doi: 10.1016/j.amj.2017.10.005. Epub 2017 Dec 6. No abstract available. PMID 29478578
- [Background] Ringburg AN, de Ronde G, Thomas SH, van Lieshout EM, Patka P, Schipper IB. Validity of helicopter emergency medical services dispatch criteria for traumatic injuries: a systematic review. Prehosp Emerg Care. 2009 Jan-Mar;13(1):28-36. doi: 10.1080/10903120802472012. PMID 19145521
- [Background] Fevang E, Lockey D, Thompson J, Lossius HM; Torpo Research Collaboration. The top five research priorities in physician-provided pre-hospital critical care: a consensus report from a European research collaboration. Scand J Trauma Resusc Emerg Med. 2011 Oct 13;19:57. doi: 10.1186/1757-7241-19-57. PMID 21996444
- [Background] Galvagno SM Jr, Sikorski R, Hirshon JM, Floccare D, Stephens C, Beecher D, Thomas S. Helicopter emergency medical services for adults with major trauma. Cochrane Database Syst Rev. 2015 Dec 15;2015(12):CD009228. doi: 10.1002/14651858.CD009228.pub3. PMID 26671262
- [Background] Scholten AC, Haagsma JA, Panneman MJ, van Beeck EF, Polinder S. Traumatic brain injury in the Netherlands: incidence, costs and disability-adjusted life years. PLoS One. 2014 Oct 24;9(10):e110905. doi: 10.1371/journal.pone.0110905. eCollection 2014. PMID 25343447
- [Background] Doucet J, Bulger E, Sanddal N, Fallat M, Bromberg W, Gestring M; Emergency Medical System Subcommittee, Committee on Trauma, American College of Surgeons. Appropriate use of helicopter emergency medical services for transport of trauma patients: guidelines from the Emergency Medical System Subcommittee, Committee on Trauma, American College of Surgeons. J Trauma Acute Care Surg. 2013 Oct;75(4):734-41. doi: 10.1097/TA.0b013e3182a5389e. No abstract available. PMID 24064891
- [Background] Rathore SS, Curtis JP, Chen J, Wang Y, Nallamothu BK, Epstein AJ, Krumholz HM; National Cardiovascular Data Registry. Association of door-to-balloon time and mortality in patients admitted to hospital with ST elevation myocardial infarction: national cohort study. BMJ. 2009 May 19;338:b1807. doi: 10.1136/bmj.b1807. PMID 19454739
- [Background] Pinto DS, Kirtane AJ, Nallamothu BK, Murphy SA, Cohen DJ, Laham RJ, Cutlip DE, Bates ER, Frederick PD, Miller DP, Carrozza JP Jr, Antman EM, Cannon CP, Gibson CM. Hospital delays in reperfusion for ST-elevation myocardial infarction: implications when selecting a reperfusion strategy. Circulation. 2006 Nov 7;114(19):2019-25. doi: 10.1161/CIRCULATIONAHA.106.638353. Epub 2006 Oct 30. PMID 17075010
- See also: Educational programs to improve emergency care based on evidence based medicine. — http://www.naemt.org/education/education-overview